CLINICAL TRIAL: NCT04944654
Title: Efficacy, Tolerability and Acceptability of the Single Table Regimen (STR) Biktarvy® by Trans People Living With HIV (TPLWH)
Brief Title: Efficacy, Tolerability and Acceptability of Biktarvy by TPLWH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial set up was delayed, funding support no longer available
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Gilead Sciences (Industry); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRF005
Record Dates: First submitted 2021-06-14; First posted 2021-06-29 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Open label, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned intervention (Experimental): Biktarvy OD for 96 weeks
  Interventions: Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet

INTERVENTIONS:
Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet — Combination single tablet anti-retroviral therapy: bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg

SUMMARY:
This is a clinical trial for TPLWH (Trans People Living with HIV) who are stable on cART with an undetectable viral load or a detectable viral load but no resistance to NRTIs and InSTI. Following written consent and screening procedures, study subjects will undergo a switch (or will restart) of their combination antiretroviral therapy (cART) to Biktarvy. The goal of this research project is to recruit an understudied population into a controlled clinical trial aimed at optimizing TPLWH cART. This will be demonstrated by measuring viral load outcomes at regular intervals, with a focus on viral load results 48 weeks after Biktarvy initiation (primary outcome).

DETAILED DESCRIPTION:
The goal of this research project is to recruit an understudied population into a controlled clinical trial aimed at optimizing TPLWH cART. This will be demonstrated by measuring viral load outcomes at regular intervals, with a focus on viral load results 48 weeks after Biktarvy initiation (primary outcome). A series of secondary endpoints will also be investigated to further demonstrate the benefits of Biktarvy use in a population that is known to experience a number of factors that correlate to poor cART adherence, higher viral loads, and worst clinical outcome.

This study is an Open-label, single arm, phase IV, multi-centre TPLWH who are stable on cART with an undetectable viral load or a detectable viral load but no resistance to NRTIs and InSTI. Each participant will act as his / her own control. The study duration is 96 weeks (primary endpoint will be at 48 weeks).

Screening and Baseline visit (Day 1):

Demographics, medical history and concomitant medications (CMs) review Physical examination, height, weight, waist circumference, vital signs (including temperature, blood pressure, heart rate and respiratory rate) Review of inclusion and exclusion criteria Written informed consent cART prescription Combination antiretroviral treatment initiation (treatment should commence within 28 days after the screening visit.

Urinalysis (macro-analysis and pregnancy test ) Hepatitis B/C testing (results from samples taken up to 14 days before baseline visit can be used). Chronic hepatitis B and history of hepatitis C (cured) are allowed Blood chemistry and haematology (results from samples taken up to 14 days before baseline visit can be used) Viral load Waist circumference at baseline and week 48 Questionnaires: Pittsburgh sleep questionnaire, Wellness thermometer, Barriers to Adherence questionnaire (only at baseline, week 24, 48, 96). GAD-7 and PHQ-9 at baseline and week 48.

Metabolics/metabolomics (plasma and urine) at baseline

Follow-up visits:

Week 4 (Day 22-36) Week 12 (Day 78-92) Week 24 (Day 162-176) Week 48 (Day 330-344) Week 60 (Day 426-440) Week 72 (Day 510-524) Week 96 (Day 670-684) cART prescription (Weeks 4, 12, 24, 48, 60, 72, and 96) Vital signs Weight, waist circumference Blood chemistry and haematology at local laboratory (see appendix 1) Urinalysis Viral load, CD4/CD8 counts (only at weeks 48 and 96 at local laboratory) Questionnaires: Pittsburgh sleep questionnaire, Wellness thermometer, Barriers to Adherence questionnaire (only at weeks 24, 48, 96). GAD-7 and PHQ-9 at baseline and week 48.

Concomitant medication check and adverse events review Metabolic and/or metabolomics changes (plasma and urine) following the switch to Biktarvy at weeks 24, 48 and 96.

Waist circumference at baseline and week 48

End of study visit (within 30 days after End of Treatment) OR Early Termination Visit (within 30 days of premature withdrawal) Vital signs Viral Load Blood chemistry and haematology Urinalysis Concomitant medication check and adverse events review

ELIGIBILITY:
Inclusion Criteria:

* Participant self-identifies as transgender and/or has a current gender identity which differs from gender assigned at birth (includes all gender diverse people)
* Age > 18 years
* HIV infection diagnosis at any time before study consent
* Willing to sign an informed consent and take part in the study
* On an antiretroviral regimen with an undetectable viral load or off an antiretroviral regimen with a detectable viral load (the cART can have been stopped for any clinical or personal reason; if on cART with a detectable viral load and no resistance to any of the component of Biktarvy, the patient is also eligible.
* A female may be eligible to enter and participate in the study if she:

  * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * is of child-bearing potential with a negative pregnancy test at Screening (& baseline visit) and agrees to use one of the methods of contraception to avoid pregnancy indicated during the study and for a period of 12 weeks after the study.
  * Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 3) must be using an adequate method of contraception as listed the Protocol to avoid pregnancy in their partner throughout the study and for a period of at least 12 weeks after the study.

Exclusion Criteria:

* Age < 18 years
* Unable to take part in the study according to the Investigator opinion (example: unable to understand the study information leaflet, unable to provide written consent, etc.)
* History of virological failure while on a cART containing NRTIs and InSTIs and development of resistance to NRTIs and InSTI
* Use of medications that are known to interact with Biktarvy. Contraindications given in appendix 4 and full information on drug-drug interactions given in SmPC.
* Hypersensitivity to active substance or excipient of Biktarvy as listed in SmPC.
* Women planning pregnancy or who are pregnant or breast feeding.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical or anal intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject prior to randomisation.
* Known acute or chronic viral hepatitis including, but not limited to, A, B, or C. Chronic hepatitis B and history of hepatitis C (cured) are allowed
* Any investigational drug within 30 days prior to the trial drug administration
* Any other condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 1 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Measure of viral load | 48 weeks
  Proportion of subject with HIV viral load < 50 copies/mL from baseline to week 48

SECONDARY OUTCOMES:
Measure of viral load | week 96
  Proportion of subject with HIV viral load < 50 copies/mL from baseline to week 24 and 96.
Change in clinical outcomes | week 96
  Occurrence of changes in clinical outcomes such as bone health, kidney function, cardiovascular risk, BMD, weight, BMI.
Drug-drug interactions | week 96
  To evaluate the potential for drug-drug interactions in TPLWH who switch from their cART to Biktarvy® based on the University of Liverpool Drug interaction website or other sources of drug interaction knowledge, including prescribed drugs, hormones, over the counter medications and recreational drugs.
Changes in CD4 count and CD4:CD8 ratio | week 48 and 96
  Changes in CD4 count and CD4:CD8 ratio during the course of the study
Patient questionnaires | week 24, 48 and 96
  Patient reported outcomes will be collected following the administration of specific questionnaires (including Wellness thermometer, sleep questionnaire, barriers to adherence questionnaire) in relation to the drug switch) at baseline and weeks 24, 48 and 96.Questionnaire such as GAD-7 and PHQ-9 will also be administered at baseline and at week 48.
Measurement of waist circumference | week 48
  To assess change in waist circumference at baseline and week 48.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — Chelsea and Westminster Hospital NHS Foundation Trust, London
Locations (1):
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No